CLINICAL TRIAL: NCT00184639
Title: Comparison of Efficacy and Safety of Insulin Detemir and Insulin Semilente®MC in Children, Adolescents and Young Adults With Type 1 Diabetes on Basal-Bolus Regimen.
Brief Title: Comparison of Insulin Detemir and Insulin Semilente®MC in Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1630
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir

SUMMARY:
This trial is conducted in Europe.

A 32-week efficacy and safety comparison of insulin detemir and insulin semilente MC in children between 6 and 21 years with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Current intensified insulin treatment
* Injection of insulin Semilente®MC at bedtime for at least 6 weeks
* BMI maximum 32 kg/m^2
* HbA1c > 5.5 % and < 12.0 %

Exclusion Criteria:

* Current treatment with premixed insulin(s)
* Impaired hepatic or renal function
* Recurrent major hypoglycaemia

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2004-08-16 (Actual); Primary Completion 2005-11-22 (Actual); Study Completion 2005-11-22 (Actual)

PRIMARY OUTCOMES:
Fasting plasma glucose | after 16 and 32 weeks, respectively

SECONDARY OUTCOMES:
Adverse events
HbA1c results at the end of each treatment period
Blood glucose
Standard Laboratory Safety Parameters
Hypoglycaemia

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Germany (2):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Hanover

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com